CLINICAL TRIAL: NCT00247689
Title: Methylphenidate Studies for Drug Abuse Vulnerability Molecular Genentics
Status: Terminated | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905381; 05-DA-N381
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2015-02-27

CONDITIONS: Substance Abuse
Keywords: Ritalin; Substance Abuse; Allelic Variants; Genotype; Addiction-Associated Human Gene Variants; Methylphenidate
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Research has shown that several human genes have been associated with vulnerability to substance abuse and dependence. However, little is known about how people with these genetic tendencies react to drugs in controlled settings.
* Methylphenidate, also known as Ritalin, is commonly prescribed for a number of conditions, including attention deficit disorder. Because methylphenidate is widely used in studies of brain chemistry and behavior and has relatively low risks associated with it use, researchers are interested in seeing how it affects the thinking processes of people with apparent genetic vulnerability to drug abuse.

Objectives:

- To evaluate whether individuals with apparent genetic vulnerability to drug abuse react differently to methylphenidate than people who do not have this vulnerability.

Eligibility:

- Individuals at least 18 years of age or older who have participated in the NIDA protocol Allelic Linkage in Substance Abuse.

Design:

* Participants will be asked to avoid using a number of over-the-counter medications, including antihistamines, cough medicines, and nasal decongestants, for 24 hours before the study day. Participants will also be asked to avoid consuming caffeinated beverages, nicotine or tobacco products, or alcohol on the morning of the day of the study, and will provide a urine sample at the start of the study to be tested for chemicals that may interfere with the study.
* Because of the nature of the study drug, participants will not be allowed to drive to the clinical center on the day of the study. (Return transportation will be arranged.)
* At the start of the study, participants will take two tablets (each 1 hour apart), and will not be told whether the tablets are the study drug or a placebo.
* Participants will give regular answers to questions about mood and thinking processes on a computer for approximately 5 hours. Blood samples will be taken during this part of the study.

DETAILED DESCRIPTION:
Scientific Goals. We and others have now identified several human chromosomal regions that contain genetic markers that have been associated with vulnerability to substance abuse/dependence in several different human populations (Uhl et al, 2002). However, little is known about the biological or behavioral mechanisms by which specific molecular genetic characteristics enhance risks for drug disorders. This protocol will test hypotheses that genetically-mediated individual differences in acute responses to abused substances contribute to the mechanisms through which specific human allelic variants influence individual differences in vulnerability to drug abuse/dependence. This protocol will characterize individual differences in responses to oral methylphenidate (30 mg) (also known as Ritalin). We have chosen this agent due to a) its wide clinical use, b) its moderate to low risks which are largely well-understood as a result of this widespread use, and c) its prior usefulness to us and others as a probe for reward system activities in, for example, patients with dopaminergic brain lesions (Persico et al 1998). We have chosen this dose due to: a) our prior success with this dose, even in a brain lesioned clinical population (Persico et al 1998) b) our preliminary work with candidate gene studies in individuals administered oral doses of up to 60-70 mg (GRU et al, in preparation) c) consultations with other workers in the field who advise use of this dose and who have used doses of 0.5 mg/kg intravenously in prior work with few reported adverse events (Volkow et al, 2003).

We will study individuals who are selected based on their genotypes. We will test the hypothesis that individuals who display combinations of the abuse-associated and/or resistance-associated allelic variants at different genomic loci that we and others have reproducibly associated with substance abuse (Uhl et al 2002) will differ in their acute responses to methylphenidate administration. We will also perform exploratory analyses of these data. We will study the genotypes of individuals who display high- or low-level responses to oral methylphenidate administration. Both the hypothesis-testing and exploratory aspects of this study will allow us to identify which addiction-associated human gene variants can alter subjective and physiologic responses to administration of methylphenidate.

Method. We will study previous participants in study #148 (90-DA-N448) who have already consented to recontact from NIDA personnel. We will select individuals who are eligible for study participation based on their genotypes at markers whose alleles differ between drug abusers (those who report significant lifetime use and dependence on at least one illegal substance) and controls (individuals free from significant lifetime use of any addictive substances) as well as allelic variants in genes expressed in reward circuits. Patients will receive psychiatric and medical screening. Eligible volunteering participants will have a one-day study session in which they receive oral placebo and oral methylphenidate (30 mg) in single-blinded fashion. This design was chosen to allow study participation by a larger fraction of eligible participants than those likely to consent to inpatient stays and longer designs. Subjective methylphenidate effects, plasma levels of methylphenidate and heart rate will be assessed periodically before and for 4 hours after the drug is administered. Methylphenidate was chosen as a probe because: (1) its mechanism of action directly involves central monoaminergic reward pathways, including dopamine and norepinephrine transporter inhibition, (2) there is such broad clinical experience with the drug that significant side effects are well known to be of low frequency in broad populations (3) there are individual differences in methylphenidate subjective responses documented in several sorts of studies, including the studies of Parkinsonian patients and controls previously reported from our group.

Hypothesis. We advance a two-tailed hypothesis that subjective liking VAS responses to methylphenidate will be different in those individuals with multiple candidate genetic characteristics that are related to enhanced vulnerability to substance abuse/dependence compared to matched controls with few of these genomic characteristics. Confidence will be greatest for those associations that are consistent among both Caucasian/European American and African American participants, an internal replication built into this design.

Benefits. The results will have important implications for possible mechanisms by which genetic vulnerability to substance abuse (particularly psychostimulants) is expressed in humans. The findings will also bear on genetic predictors of the response to methylphenidate, which may be important for attention deficit hyperactivity disorder, narcolepsy and other clinical disorders in which drugs of this class are used therapeutically.

Risks. Methylphenidate is also known as Ritalin, and is commonly prescribed for a number of clinical conditions including attention deficit/hyperactivity syndrome. The drug has been used for many individuals with few serious complications. Individuals who use this drug for long periods of time may show nervousness and sleep changes. Skin rashes, appetite suppression, nausea, dizziness, heart palpitations, pulse and heart rhythm changes, headache, abnormal movements, sleepiness, chest pain, abdominal pain, liver function changes, blood cell changes and changes in thinking have also been rarely reported in individuals who use this drug chronically. A review of patients taking a treatment dose of methylphenidate for ADHD revealed serious cardiovascular adverse events in patients with underlying serious heart problems or defects, and reports of stroke and heart attack in adults with certain risk factors, (i.e. untreated high blood pressure and a history of coronary artery disease). Another review of patients taking a treatment dose of methylphenidate for ADHD revealed a slight increased risk (about 1 per 1,000) for drug-related psychiatric adverse events, such as hearing voices, becoming suspicious for no reason, or becoming manic, even in patients who did not have previous psychiatric problems. Additional modest to minimal risks to participants include the risks of venous catheterization and blood withdrawal, including pain, bruising and bleeding, and the risks of confidentiality. We will minimize each of these more than minimal risks by appropriate exclusionary criteria, medical screening, use of low/moderate drug doses, evaluation prior to discharge, availability of taxi for return home, aseptic methods, small total amounts of blood drawn, standard minimal risk recording procedures, coded, locked data and Confidentiality Certification of this work.

ELIGIBILITY:
* INCLUSION CRITERIA:

Self-reported White/Caucasian or Black/African American individual who have participated in the protocol #148 (90-DA-N448) in order to obtain the molecular genetic variables needed in the current study. We will contact only those individuals (substance abusers, non-substance abusing controls, and family members if the proband does not qualify) who have participated in study #148 (90-DA-N448) at times when their consent included written agreement to be contacted at a later date and are enrolled at the NIDA Intramural Research Program.

EXCLUSION CRITERIA:

1. Do NOT have a history of

   1. Seizures,
   2. Head injury resulting in unconsciousness and/or requiring hospitalization
   3. Cardiovascular abnormalities (i.e. murmur)
   4. Uncontrolled or untreated hypertension

      -Diastolic >95 mmHg and/or Systolic > 145 mmHg
   5. Clinically significant anxiety, depression, and/or panic disorder
   6. Coronary artery disease.

      History of known coronary artery disease,
      * History of a prior myocardial infarction or stroke.
      * An 12 lead EKG will be done during screening (no more than three months prior to enrollment), reviewed by an M.D, and may be sent to an outside cardiologist for manual reading.
      * EKG abnormalities which will EXCLUDE a subject will include the following: QTc interval > 450 ms or changes suggesting acute ischemia, second or third degree heart block, left bundle branch block, atrial fibrillation, signs of left ventricular hypertrophy or other clinically important arrhythmias.
   7. Dependence on methylphenidate or a psychostimulant
   8. History of an adverse reaction to cocaine, methylphenidate, amphetamine, other psychostimulant, herb and/or over the counter medication
   9. Urine sample positive for a psychostimulant on the day of the study. (An observed urine specimen will be tested on the day of the study)
   10. Clinically significant abnormal renal and/or liver function

       * Renal (lab cut off ): BUN > 35mg/dl; Cr > 2.0 mg/dl
       * Liver (lab cut off): AST > 200 U/L; ALT >200 U/L; Alk P > 200 U/L; GGT> 400 U/L
   11. Diagnosed with a movement disorder
   12. Diagnosed with glaucoma
   13. Currently taking any of the following: monoamine oxidase inhibitors (within 2 weeks of protocol participation), insulin, and/or a psychostimulant
   14. A major medical diagnosis (i.e. .stroke, rheumatoid arthritis on therapy, diabetes)
2. Competent to give informed consent. Competency of research participation at the NIDA will be determined by a Shipley Institute of Living Scales estimated IQ score of 80 or greater and an SCL-90-R Global Severity Index T-score of 70 or less. Cognitive impairment will be defined using the Shipley Institute of Living Scale or WRAT (equivalent to WAIS-R IQ < 79). With individuals having SCL-90-R scores greater than 70 referred for evaluation to a Counselor or Physician before admission to the study can be complete. The counselor or physician using his/her clinical judgment will make 1 of 2 determinations: a) The applicant may continue with the screening process; b) The applicant is disqualified from participation in the study and an appropriate referral is made if indicated.
3. To evaluate the understanding of the study, its risk and benefits, and how to withdrawal from the study at anytime will be determined by a Consent Quiz score of 80 percent or greater (answering 8 of 10 questions correctly) in NIDA participants

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2004-12-22; Study Completion 2015-02-27

CONTACTS AND LOCATIONS:
Overall Officials: George R Uhl, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Background] Brown WA, Corriveau DP, Ebert MH. Acute psychologic and neuroendocrine effects of dextroamphetamine and methylphenidate. Psychopharmacology (Berl). 1978 Jul 6;58(2):189-95. doi: 10.1007/BF00426906. No abstract available. PMID 98790
- [Background] Clark CR, Geffen GM, Geffen LB. Catecholamines and attention. II: Pharmacological studies in normal humans. Neurosci Biobehav Rev. 1987 Winter;11(4):353-64. doi: 10.1016/s0149-7634(87)80007-6. PMID 3325865
- [Background] Evans WE, McLeod HL. Pharmacogenomics--drug disposition, drug targets, and side effects. N Engl J Med. 2003 Feb 6;348(6):538-49. doi: 10.1056/NEJMra020526. No abstract available. PMID 12571262